CLINICAL TRIAL: NCT06914921
Title: "A Non-Inferiority Randomized Controlled Trial of Enteric-Coated Peppermint Oil Versus Standard Antispasmodic in SLC6A4 (5-HTTLPR) Carriers With Irritable Bowel Syndrome."
Brief Title: Enteric-Coated Peppermint Oil Versus Standard Antispasmodic in SLC6A4 (5-HTTLPR) Carriers With Irritable Bowel Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Center for New Medical Technologies, Novosibirsk, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SW027
Record Dates: First submitted 2025-04-04; First posted 2025-04-07 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: supplements; genetics; peppermint oil
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — peppermint oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enteric-coated peppermint oil capsules (~180 mg total peppermint oil/ capsule) to ensure release in (Experimental)
  Interventions: Dietary Supplement: Peppermint Oil
- A standard antispasmodiс (Active Comparator): A standard antispasmodic (e.g., mebeverine 135 mg).
  Interventions: Drug: A standard antispasmodic

INTERVENTIONS:
Dietary Supplement: Peppermint Oil — Enteric-coated peppermint oil capsules (~180 mg total peppermint oil/ capsule) to ensure release in the small intestine.
  1 capsule three times daily, 30 minutes before meals, for 12 weeks.
  Arms: Enteric-coated peppermint oil capsules (~180 mg total peppermint oil/ capsule) to ensure release in
Drug: A standard antispasmodic — A standard antispasmodic (e.g., mebeverine 135 mg). 1 tablet three times daily, before meals, for 12 weeks.
  Arms: A standard antispasmodiс

SUMMARY:
This study is a non-inferiority, double-blind, randomized controlled trial comparing enteric-coated peppermint oil with a standard antispasmodic (e.g., mebeverine) in adult IBS patients who carry at least one "S" allele in the SLC6A4 (5-HTTLPR) polymorphism. The primary goal is to see whether peppermint oil provides symptom relief (measured by IBS severity scores) that is not worse than the antispasmodic by more than a predefined margin (30 points on the IBS-SSS). Secondary goals include evaluating differences in abdominal pain, stool patterns, quality of life, and adverse event profiles, with a focus on peppermint oil's tolerability. About 224 participants (112 per arm) will be enrolled, with allowances for dropout, to detect non-inferiority at 80% power. After 12 weeks of treatment, results will inform whether peppermint oil is a viable, well-tolerated alternative to standard antispasmodics, especially in patients with heightened GI sensitivity linked to the SLC6A4 polymorphism.

DETAILED DESCRIPTION:
This double-blind, parallel-group, non-inferiority RCT will randomize ~250 adults (18-65 y) who meet Rome IV criteria for IBS and carry at least one short 5-HTTLPR (SLC6A4) allele to enteric-coated peppermint-oil capsules (180 mg three times daily) or the standard antispasmodic mebeverine (135 mg three times daily) for 12 weeks. Because the S-allele reduces serotonin-transporter expression and heightens visceral sensitivity, the study targets a genetically defined subgroup in which menthol's smooth-muscle-relaxing calcium-channel blockade may yield clinically meaningful benefit with fewer anticholinergic effects. Randomisation (1 : 1) is web-based, stratified by genotype and centre, and treatments are packaged identically to maintain blinding of participants, investigators, and outcome assessors. The primary endpoint is change from baseline in the IBS Severity Scoring System at week 12; non-inferiority is met if the upper bound of the two-sided 95 % CI for the treatment difference (peppermint - mebeverine) is ≤ +30 points. A mixed-model repeated-measures analysis will be applied to both intention-to-treat and per-protocol populations, providing 80 % power with ~112 evaluable patients per arm. Secondary outcomes include abdominal-pain intensity, stool form, quality of life, global satisfaction, and adverse events; safety is tracked via weekly contacts, laboratory tests, and an independent data-safety monitoring board. Demonstrating that peppermint oil is at least as effective as mebeverine while better tolerated would support its use as a genotype-guided first-line therapy for IBS.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years.
* Diagnosis of Irritable Bowel Syndrome by Rome IV criteria, with at least moderate severity (IBS-SSS ≥ 175).
* SLC6A4 genotyping confirms at least one S allele (SS or SL).
* Able and willing to provide informed consent and comply with study procedures.

Exclusion Criteria:

* L/L genotype of 5-HTTLPR.
* Known organic GI diseases (e.g., IBD, celiac disease).
* Severe/unstable comorbidities (e.g., cardiac, hepatic, or renal dysfunction).
* Use of peppermint oil, antispasmodics, or investigational drugs within 30 days prior to enrollment.
* . Known hypersensitivity to peppermint or mebeverine.
* Pregnancy or breastfeeding.
* Significant psychiatric illness that, in the investigator's judgment, might interfere with participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2024-02-04 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome | 12 weeks
  Symptom severity in this trial is captured with the IBS-SSS (IBS Severity Scoring System): 0 = no symptoms to 500 = most severe symptoms

SECONDARY OUTCOMES:
Numeric Rating Scale (for abdominal pain) | 12 weeks
  Range: 0 = no pain to 10 = worst imaginable pain
Abdominal Pain: Measured by visual analog score | 12 weeks
  0 as a minimum value and 10 maximum value
Stool Consistency: Bristol Stool Form Scale | 12 weeks
  range 1-7, 1 = separate hard lumps/constipation, 7 = watery stool/diarrhea; higher scores indicate looser stool
Quality of Life: Irritable Bowel Syndrome Quality of Life Questionnaire | 12 weeks
  transformed score 0-100; higher scores indicate better IBS-specific quality of life
Quality of Life: 36-Item Short Form Health Survey | 12 weeks
  domain and summary scores 0-100; higher scores indicate better health-related quality of life
Adverse Events: Incidence | 12 weeks
  Number of any adverse events
Global Patient Satisfaction: Five-point Likert Scale | 12 weeks
  ange 1-5 (1 = very dissatisfied, 5 = very satisfied); higher scores indicate greater satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Center for New Medical Technologirs, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No